CLINICAL TRIAL: NCT02075086
Title: Angiogenic Switch as Predictor of Response to Chemotherapy in Patients With Metastatic Colorectal Cancer
Brief Title: Angiogenic Switch in Patients With Colorectal Cancer
Acronym: ANGIOSWITCH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Hospital de Madrid (Other)
Responsible Party: Principal Investigator, Sofia Perea, Director Clinical Trials Unit., MD, PhD, Grupo Hospital de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANGIOSWITCH2011
Record Dates: First submitted 2011-11-17; First posted 2014-03-03 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer
Keywords: angiogenic switch; plasma cytokines; Colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy treatment (Experimental): Chemotherapy treatment with Xelox or Xeliri and bevacizumab
  Interventions: Drug: Xelox or Xeliri Bevacizumab

INTERVENTIONS:
Drug: Xelox or Xeliri Bevacizumab — Chemotherapy treatment
  Other Names: Cytokines measure; Angiogenic study

SUMMARY:
A group of colorectal cancer (CRC) patients treated with chemotherapy and Bevacizumab (Bev) maintain the same sensitivity after progression to maintenance treatment because they remain dependent on VEGF angiogenic mediator, while other patients in whom there is an angiogenic switch (AS) become dependent on other angiogenic cytokines and become resistant to Bev chemotherapy combinations .

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV colorectal adenocarcinoma.
* Age ≥ 18 years .
* Measurable disease by RECIST criteria.
* Life expectancy ≥ 6 months.
* Candidate to receive treatment with first-line chemotherapy.
* Availability of tumor tissue.

Exclusion Criteria:

* Patients who have received prior treatment with first-line chemotherapy for metastatic disease.
* Patients in whom there is contraindication to the administration of either drug used in the study: capecitabine, irinotecan, oxaliplatin or Bev.
* Patients receiving anticoagulant oral treatment.
* Patient with diagnosis of other malignancies within 5 years prior to diagnosis except basal cell carcinoma or cervical carcinoma · in situ. · The inclusion of patients with malignant disease diagnosed more than 5 years ago without recurrence in the previous 3 years will be analyzed individually
* Patients with bone disease as the only manifestation of the disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  Days from cycle one day one to progression

SECONDARY OUTCOMES:
Feasibility | 2 years
  Feasibility of doing a clinical prospective trial with a measure od plasma citoquines.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cubillo, MD PhaD, Principal Investigator — Grupo Hospital de Madrid
Locations (1):
- Centro Integral oncológico Clara Campal, Madrid, Spain